CLINICAL TRIAL: NCT04828590
Title: Assessment of the DiAgnostic Performance of DeepVessel FFR in SuspecTed Coronary Artery Disease
Brief Title: The ADAPT Study: Assessment of the DiAgnostic Performance of DeepVessel FFR in SuspecTed Coronary Artery Disease
Acronym: ADAPT
Status: Completed | Type: Observational
Sponsor: Keya Medical (Industry)
Collaborators: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: DVFFR ADAPT Study
Record Dates: First submitted 2021-03-28; First posted 2021-04-02 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Patients with suspected CAD containing at least one 30%-90% coronary CTA stenosis: Patients' datasets with suspected CAD containing at least one 30%-90% coronary CTA stenosis; and ICA-FFR was measured on vessels with diameters greater than 2 mm will be analyzed. Diagnostic performance based on CT-derived FFR using DVFFR software will be compared with the diagnostic performance from ICA-FFR measurements.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Due to observational study

SUMMARY:
DEEPVESSEL FFR is a medical device that is designed to extract three- dimensional coronary tree structures and generate computed tomography-derived fraction flow reserve (FFR) values from coronary CT angiogram images. The primary objective of this multi-center clinical validation study is to validate the clinical performance of DEEPVESSEL FFR in identifying patients with myocardial ischemia due to significant obstructive coronary artery diseases.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is the most common type of heart disease, and it is the leading cause of death worldwide in both men and women. CAD happens when the coronary arteries become hardened and narrowed, which is due to the buildup of cholesterol-containing deposits-plaque on the inner vessel wall. As the plaque grows, less blood can flow through the arteries due to the vessel narrowing. Decreased blood flow can then lead to chest pain (angina), shortness of breath, or even a heart attack.

Fractional flow reserve (FFR), a measure of blood flow reduction caused by vessel narrowing, is accepted as gold standard for assessing the functional significance of stenotic lesions. Multiple randomized trials have demonstrated that FFR has excellent diagnostic value in identifying functionally significant lesions and guiding coronary revascularization procedures. However, FFR is measured invasively through a pressure wire-based cardiac catheter procedure in the catheterization lab. Current guidelines recommend assessing myocardial ischemia of stable patients with CAD through non-invasive functional testing before considering invasive coronary angiography (ICA) or conducting myocardial revascularization.

DEEPVESSEL FFR (DVFFR) is a software medical device that is designed to extract three- dimensional coronary tree structures and generate computed tomography -derived FFR values from coronary CT angiogram (CTA) images. It uses deep learning neural networks that encode imaging, structural, and functional characteristics of coronary arteries and learn complex mapping between FFR values and the encoded information. The quantitative FFR analysis based on the coronary CTA images can help clinicians assess the physiological function in patients with CAD non-invasively.

The primary objective of this study is to evaluate the diagnostic performance of DVFFR software in identifying patients with significant obstructive CAD causing myocardial ischemia, using invasively measured ICA FFR as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

1. Patients' age ≥18 years;
2. Has coronary CTA images acquired by ≥64 multidetector row CT scanner, no earlier than 2016 and within 60 days of the ICA-FFR procedure;
3. Coronary CTA image shows at least one vessel segment (≥2mm diameter) with a diameter stenosis of 30%-90%;

Exclusion Criteria:

Patients with any of the following conditions at the time of CTA imaging:

1. Acute myocardial infarction;
2. Unstable angina;
3. Pulmonary edema;
4. Heart function classification level III and IV (NYHA heart function classification);
5. Implantable cardioverter defibrillator (ICD);
6. Prior percutaneous coronary intervention (PCI) or pacemaker surgery;
7. Prior coronary artery bypass grafting (CABG) surgery;
8. Prior heart valve replacement;
9. Prior history of complex congenital heart disease;
10. Prior history of cardiomyopathy;
11. BMI >35;
12. Coronary total occlusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with suspected CAD containing at least one 30%-90% coronary CTA stenosis.
Sampling Method: Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Sensitivity of DVFFR at the vessel level in identifying ischemic lesions, i.e. DVFFR value≤0.80, from coronary CTA images, using ICA-FFR measurement as a reference standard. | through study completion, an average of 1 year
  On the vessel level, if a vessel with at least one stenosis lesion with a FFR measurement less or equal to 0.80, this vessel is considered to be ischemic. A true positive on the vessel level is defined as a vessel containing at least one stenosis with DVFFR value ≤0.80 and its corresponding reference ICA-FFR value is also ≤0.80.
Specificity of DVFFR at the vessel level in identifying ischemic lesions, i.e. DVFFR value≤0.80, from coronary CTA images, using ICA-FFR measurement as a reference standard. | through study completion, an average of 1 year
  On the vessel level, if a vessel with at least one stenosis lesion with a FFR measurement less or equal to 0.80, this vessel is considered to be ischemic. A true positive on the vessel level is defined as a vessel containing at least one stenosis with DVFFR value ≤0.80 and its corresponding reference ICA-FFR value is also ≤0.80.

SECONDARY OUTCOMES:
Diagnostic accuracy, positive predictive value (PPV) and negative predictive value (NPV) of DVFFR at the vessel level | through study completion, an average of 1 year
  On the vessel lever, if a vessel with at least one stenosis lesion with a FFR measurement less or equal to 0.80, this vessel is considered to be ischemic. A true positive on the vessel level is defined as a vessel containing at least one stenosis with DVFFR value ≤0.80 and its corresponding reference ICA-FFR value is also ≤0.80.
Diagnostic performance including sensitivity, specificity, accuracy, PPV and NPV of DVFFR at the patient level | through study completion, an average of 1 year
  At the patient level, if a patient has at least one vessel that has been identified as causing ischemia, this patient is considered a patient positive for ischemia. A true positive on the patient level is defined as when a patient has at least one lesion with a DVFFR value ≤0.80 and its corresponding reference ICA-FFR is also ≤0.80.
Per-vessel Pearson correlation coefficient between DVFFR and ICA-FFR values | through study completion, an average of 1 year
  Correlation between CT-derived DVFFR values and wire-measured ICA-FFR values will be evaluated at the vessel level.
Diagnostic performance (including sensitivity, specificity, accuracy, PPV and NPV) in detecting hemodynamically significant coronary obstruction using DVFFR and coronary CTA alone, on both vessel level and patient level. | through study completion, an average of 1 year
  For coronary CTA, hemodynamically significant obstruction of a coronary artery is defined as a stenosis ≥50%. The per-patient stenosis degree will be specified as the most severe stenosis among the major epicardial artery vessels presented in coronary CTA.
Stratified analyses on different subgroups of subjects' data | through study completion, an average of 1 year
  Stratified analyses on different subgroups of subjects' data, ranging from patient demographics and disease conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Schoepf, MD, Principal Investigator — Medical University of South Carolina
Locations (10):
- United States (5):
  - Holy Cross Health, Fort Lauderdale, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Oregon Health & Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Medical University Innsbruck, Innsbruck, Austria
- Institute of Arnualt Tzanck, Nice, Saint-Laurent-du-Var, France
- Italy (2):
  - University of Ferrara, Ferrara
  - University of Milan, Milan
- National Institute of Cardiology, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No